CLINICAL TRIAL: NCT00296465
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Three Dosage Strengths of Pulsatile GnRH Administered Intravenously or Subcutaneously (Via Portable Infusion Pump) Compared to Oral Treatment With Clomiphene Citrate in Anovulatory or Oligoovulatory Infertile Females
Brief Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Three Dosage Strengths of Pulsatile GnRH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-05
Expanded Access: Available
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: InFertility
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Lutrepulse® 5mcg IV (Experimental): 5.0 mcg Pulsatile GnRH (Lutrepulse®) administered intravenously via portable infusion pump in a pulsatile fashion (every 90 minutes) for 4 weeks and oral placebo clomiphene citrate for 5 days
  Interventions: Drug: Pulsatile gonadotropin-releasing hormone (GnRH); Drug: Placebo Clomiphene Citrate
- Lutrepulse® 10 mcg IV (Experimental): 10.0 mcg Pulsatile GnRH (Lutrepulse®) administered intravenously via portable infusion pump in a pulsatile fashion (every 90 minutes) for 4 weeks and oral placebo clomiphene citrate for 5 days
  Interventions: Drug: Pulsatile gonadotropin-releasing hormone (GnRH); Drug: Placebo Clomiphene Citrate
- Lutrepulse® 20 mcg SC (Experimental): 20.0 mcg Pulsatile GnRH (Lutrepulse®) administered subcutaneously via portable infusion pump in a pulsatile fashion (every 90 minutes) for 4 weeks and oral placebo clomiphene citrate for 5 days
  Interventions: Drug: Pulsatile gonadotropin-releasing hormone (GnRH); Drug: Placebo Clomiphene Citrate
- Placebo IV (Placebo Comparator): Placebo Pulsatile GnRH (Lutrepulse®) administered intravenously via portable infusion pump in a pulsatile fashion (every 90 minutes) for 4 weeks and oral placebo clomiphene citrate for 5 days
  Interventions: Drug: Placebo Pulsatile GnRH; Drug: Placebo Clomiphene Citrate
- Placebo SC (Placebo Comparator): Placebo Pulsatile GnRH (Lutrepulse®) administered subcutaneously via portable infusion pump in a pulsatile fashion (every 90 minutes) for 4 weeks and oral placebo clomiphene citrate for 5 days
  Interventions: Drug: Placebo Pulsatile GnRH; Drug: Placebo Clomiphene Citrate
- Clomiphene Citrate/Placebo IV (Active Comparator): Oral clomiphene citrate (over encapsulated) for 5 days and Placebo Pulsatile GnRH (Lutrepulse®) administered intravenously via portable infusion pump in a pulsatile fashion (every 90 minutes) for 4 weeks
  Interventions: Drug: Clomiphene Citrate; Drug: Placebo Pulsatile GnRH
- Clomiphene Citrate / Placebo SC (Active Comparator): Oral clomiphene citrate (over encapsulated) for 5 days and Placebo Pulsatile GnRH (Lutrepulse®) administered subcutaneously via portable infusion pump in a pulsatile fashion (every 90 minutes) for 4 weeks
  Interventions: Drug: Clomiphene Citrate; Drug: Placebo Pulsatile GnRH

INTERVENTIONS:
Drug: Pulsatile gonadotropin-releasing hormone (GnRH) — Dosages as specified, administered either subcutaneously (SC) or intraveneously (IV) as specified, via portable infusion pump in a pulsatile fashion (every 90 minutes) for 4 weeks
  Other Names: Lutrepulse®
  Arms: Lutrepulse® 10 mcg IV; Lutrepulse® 20 mcg SC; Lutrepulse® 5mcg IV
Drug: Clomiphene Citrate — Oral clomiphene citrate (over encapsulated) for 5 days
  Other Names: Clomid
  Arms: Clomiphene Citrate / Placebo SC; Clomiphene Citrate/Placebo IV
Drug: Placebo Pulsatile GnRH — Administered either intravenously or subcutaneously via portable infusion pump in a pulsatile fashion (every 90 minutes) for 4 weeks
  Arms: Clomiphene Citrate / Placebo SC; Clomiphene Citrate/Placebo IV; Placebo IV; Placebo SC
Drug: Placebo Clomiphene Citrate — oral placebo clomiphene citrate for 5 days
  Arms: Lutrepulse® 10 mcg IV; Lutrepulse® 20 mcg SC; Lutrepulse® 5mcg IV; Placebo IV; Placebo SC

SUMMARY:
This study will be performed in approximately 132 women with anovulatory/oligoovulatory infertility.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled study will be performed in approximately 132 women with anovulatory/oligoovulatory infertility. The treatment duration will be approximately 4 weeks with pulsatile GnRH or placebo and 5 days with Clomiphene Citrate or placebo. All subjects will be screened based on inclusion/exclusion criteria, medical/infertility history and general safety assessments. Subjects that complete screening will be dispensed 100 mg of oral progesterone twice a day for 10 days to induce uterine bleeding. On Cycle Day 5 from the start of bleeding the subject will be randomly assigned to 1 of 7 treatment groups. All subjects will be monitored weekly throughout the 4 week treatment period for ovulation and intercourse will be timed. All subjects will be required to return to the study center for a total of 8 visits. In addition, all subjects with a confirmed clinical pregnancy will be monitored until fetal heartbeat is confirmed at approximately 5-6 weeks gestation

ELIGIBILITY:
Inclusion Criteria

1. Females between the ages of 18 (or 19 in the State of Alabama) and 40 years.
2. Infertile due to ovulatory dysfunction as described below:
3. Positive progesterone withdrawal test following the screening visit.
4. TSH (thyroid-stimulating hormone) levels within normal limits for the clinical laboratory or considered not clinically significant (eg, secondary to exogenous thyroid medication) by the investigator
5. Normal insulin sensitivity assessed as ratio of fasting blood glucose to fasting insulin > 4.5 at Screening
6. Male partner with recent (within 6 months prior to screening) semen analysis showing normalcy according to the local laboratory normal criteria. If screening semen analysis is borderline, the couple will be accepted into the study only if a second sample obtained prior to screening is adequate.
7. Presence of both ovaries, without evidence of clinically significant abnormality, as detected by transvaginal ultrasound
8. Normal transvaginal ultrasound with respect to uterus and adnexa (eg, no hydrosalpinx)
9. Hysterosalpingography or hysteroscopy or sonohysterogram documenting a uterine cavity consistent with expected normal function and patency of the fallopian tubes within the previous 3 years prior to screening (within 1 year prior to screening there should be no pelvic infection, endometriosis or pelvic surgery).
10. Negative serum pregnancy test (qualitative) prior to the progesterone test
11. Desire to become pregnant

Exclusion Criteria

1. Requires donor oocytes or sperm
2. Previous and current use of infertility modifiers, including insulin-sensitizing drugs
3. Primary amenorrhea/hypogonadotropic hypogonadism (eg, isolated gonadotropin deficiency or evidence of primary/premature ovarian failure)
4. Presence of any clinically relevant systemic disease (eg, diabetes mellitus, pituitary tumor, anorexia nervosa).
5. Surgical or medical condition which in the judgment of the Investigator or Sponsor may interfere with absorption, distribution, metabolism, or excretion of the drugs to be used.
6. Any pregnancy within last 3 months prior to Screening.
7. Patients with a body mass index (BMI) >30 at time of Screening
8. Total testosterone and DHEA-S >1.5 times the upper limits of normal laboratory range and prolactin > 20 ng/mL
9. Presence of abnormal uterine bleeding of undetermined origin.
10. Active or prior history of substance abuse
11. History of chemotherapy (except for gestational conditions) or radiotherapy
12. Currently breast feeding, pregnant or contraindication to pregnancy
13. Refusal or inability to comply with the requirements of the Protocol for any reason, including scheduled clinic visits and laboratory tests.
14. Documented intolerance or allergy to any of the medications used including the study medication
15. Participation in any experimental drug study within 60 days prior to Screening

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2005-02; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | Day 16

SECONDARY OUTCOMES:
Adverse events, including ovarian hyperstimulation syndrome (OHSS) | Day 1 to week 5

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Southern Fertility Center and Clinical Research, Metairie, Louisiana, United States